CLINICAL TRIAL: NCT00249535
Title: Vouchers vs. Prizes for Cocaine-Dependent Methadone Patients
Brief Title: Vouchers vs. Prizes for Cocaine-Dependent Methadone Patients - 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-13444-2; R01DA013444 (NIH)
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Cocaine Dependence
Keywords: Substance Abuse; Contingency Management
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): standard treatment plus usual magnitude prize CM
  Interventions: Behavioral: Contingency management
- 2 (Experimental): standard treatment plus higher magnitude prize CM
  Interventions: Behavioral: Contingency management
- 3 (Experimental): standard treatment plus voucher CM
  Interventions: Behavioral: Contingency management

INTERVENTIONS:
Behavioral: Contingency management — Rewards (prizes) for abstinence

SUMMARY:
The purpose of this study is to compare voucher-based contingency management (CM) procedures to a lower-cost CM system that provides opportunities to win prizes. Cocaine-dependent outpatients are randomly assigned to (a) standard treatment, (b) standard treatment plus usual magnitude prize CM, (c) standard treatment plus higher magnitude prize CM, or (d) standard treatment plus voucher CM. Urine and breath samples are collected 2-3x/week for 14 weeks. Follow-up interviews are conducted at 1,3,6 and 9 months following intake during which substance use and psychosocial functioning are assessed.

ELIGIBILITY:
Inclusion criteria:

* age > 18 years
* current DSM-IV diagnosis of cocaine dependence
* received methadone treatment at the clinic for at least 3 months
* on a stable dose of methadone (no changes in dosing) for at least one month and not presently requesting a dose alteration
* submitted one or more clinic-collected cocaine positive urine samples in the previous 3 months
* English speaking
* pass a brief quiz related to understanding of the informed consent form

Exclusion criteria:

* have a serious, uncontrolled psychiatric illness (e.g., acute schizophrenia, bipolar disorder, severe or psychotic major depression, or suicide risk)
* have dementia (<23 on the Mini Mental State Exam; Folstein et al. 1975)
* are in recovery from pathological gambling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2005-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Cocaine use | baseline and each follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Petry, Ph.D., Principal Investigator — UConn Health
Locations (1):
- UConn Health Center, Farmington, Connecticut, United States